CLINICAL TRIAL: NCT00717054
Title: A Randomized, Double-blind Comparison of Oral Aprepitant Alone vs Oral Aprepitant and Transdermal Scopolamine for Preventing Postoperative Nausea and Vomiting
Brief Title: Comparison of Aprepitant Versus Aprepitant and Transdermal Scopolamine for Preventing Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00659737
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-09

CONDITIONS: Nausea; Vomiting
Keywords: postoperative nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting | interventions — Aprepitant; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant and Scopolamine group (Active Comparator): Patients receive aprepitant and scopolamine for prevention of postoperative nausea and vomiting then were followed through the post operative period looking for nausea, vomiting, composite, and rescue medication utilization. This was compared to patients receiving aprepitant and scopolamine placebo looking for a difference in incidence of events.
  Interventions: Drug: Aprepitant; Drug: Scopolamine
- Aprepitant and Scopolamine Placebo Group (Placebo Comparator): Patients receiving aprepitant and placebo scopolamine for prevention of postoperative nausea and vomiting then followed through the post operative period looking for signs of nausea, vomiting, composite, and rescue medication utilization. This was compared to patients receiving aprepitant and scopolamine looking for a difference in incidence of events.
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Aprepitant — Aprepitant 40mg PO one time at least one hour prior to induction of anesthesia
  Other Names: Emend
  Arms: Aprepitant and Scopolamine group
Drug: Scopolamine — Scopolamine transdermal applied to skin behind the ear one hour prior to surgery
  Other Names: Scopace; Transdermal scopolamine

SUMMARY:
The purpose of this study is to compare the incidence of nausea, vomiting, need for rescue medication, prolonged PACU time, and unplanned hospital admission in patients with high risk for post-operative nausea and vomiting (PONV) treated with oral aprepitant with or without transdermal scopolamine preoperatively.

DETAILED DESCRIPTION:
Aprepitant, a selective antagonist of neurokinin-1 (NK-1) receptors, blocks the emetic effects of substance P. NK-1 receptors are found on vagal afferents in the gastrointestinal tract and in the nucleus tractus solitaries in the brain. Substance P action on the NK-1 receptors in the central nervous system (CNS) is one of the final pathways to an emetic response.

Scopolamine antagonizes muscarinic type 1 (M1) and histamine type 1 (H1) receptors in the CNS, hypothalamus, and vomiting center. The noradrenergic system is also suppressed resulting in a diminished response to vestibular stimulation. Surgical procedures, opioids, and movement postoperatively all stimulate the vestibular system making scopolamine effective prophylaxis for PONV.

In adults undergoing general anesthesia with inhalational anesthetic agents, predictive risk factors for PONV include female sex, history of PONV or motion sickness, nonsmoking status, and the use of postoperative opioids. The frequency of PONV is 10% with zero, 21% with one, 39% with two, 61% with three, and 79% with 4 risk factors. The type of surgery also plays a major role. High risk procedures include intrabdominal, laparoscopic, orthopedic, major gynecologic, thyroid, otolaryngological, neurosurgical, breast, and plastic surgery.

Improving PONV prophylaxis would have a profound impact on patient care. Decreasing the incidence of nausea, vomiting, need for rescue medication, prolonged PACU time, and unplanned admissions is beneficial. Recent evidence suggests multiple drug therapy is superior to single agents. The correct preoperative treatment medication is instrumental in the outcome. This study compares the incidence of nausea, vomiting, need for rescue medication, prolonged PACU time, and unplanned hospital admission in patients with high risk for PONV treated with oral aprepitant with or without transdermal scopolamine preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* American Society of Anesthesiology (ASA) physical status 1-3
* If on oral contraceptive, must be willing to use back up method for 1 month
* Must have 2 risk factors for PONV

Exclusion Criteria:

* History of vomiting due to middle ear infection, nervous system disorder, or other condition
* Procedure less than 1 hour
* Pregnant or breast feeding
* Antiemetic medication in previous 24 hours
* Narrow-angle glaucoma
* Allergic to belladonna alkaloids
* Hypersensitive to barbiturates
* Prostate hypertrophy
* Severe hepatic disease
* On chemotherapy taking aprepitant
* Fever
* Sepsis
* Taking any of the following medications: Orap, Seldane, Hismanal, Propulsid, Phenytoin, Phenothiazines, Tricyclic antidepressants, Meperidine, Tolbutamide, Aluminum and Magnesium containing Antacids, Anti-cholinergics, Coumadin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Green, DO, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant and Placebo Scopolamine Group: Patients receiving aprepitant and placebo scopolamine for prevention of postoperative nausea and vomiting then followed through the post operative period looking for signs of nausea, vomiting, composite, and rescue medication utilization. This was compared to patients receiving aprepitant and scopolamine looking for a difference in incidence of events.
  Aprepitant: Aprepitant 40mg PO one time at least one hour prior to induction of anesthesia
  Scopolamine: Placebo Scopolamine transdermal applied to skin behind the ear one hour prior to surgery
Period: Overall Study
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Placebo Scopolamine Group
Started | 58 | 57
Completed | 58 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Placebo Scopolamine Group | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.06) | 47.2 (11.27) | 46.8 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nausea and Vomiting
Time Frame: 24 hours postoperatively
Measure: Number; unit: participants
Groups:
- Aprepitant and Placebo Scopolamine Group: Patients receiving aprepitant and placebo scopolamine for prevention of postoperative nausea and vomiting then followed through the post operative period looking for signs of nausea, vomiting, composite, and rescue medication utilization. This was compared to patients receiving aprepitant and scopolamine looking for a difference in incidence of events.
  Aprepitant: Aprepitant 40mg PO one time at least one hour prior to induction of anesthesia
  Placebo Scopolamine: Placebo Scopolamine transdermal applied to skin behind the ear one hour prior to surgery
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Placebo Scopolamine Group
Number analyzed (Participants) | 58 | 57
participants | 24 | 29

2. Secondary Outcome: Number of Participants With Nausea and Vomiting in PACU
Time Frame: Postoperatively, up to 2 hours
Measure: Number; unit: participants
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Placebo Scopolamine Group
Number analyzed (Participants) | 58 | 57
participants | 35 | 39

3. Secondary Outcome: Total Vomiting
Time Frame: 24 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Scopolamine Placebo Group
Number analyzed (Participants) | 58 | 57
participants | 5 | 2

4. Secondary Outcome: Need for Antiemetic Medication
Time Frame: 24 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Scopolamine Placebo Group
Number analyzed (Participants) | 58 | 57
participants | 23 | 21

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aprepitant and Scopolamine Group | Aprepitant and Scopolamine Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 34/58 | 29/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant and Scopolamine Group (N=58) | Aprepitant and Scopolamine Placebo Group (N=57)
Dry mouth (General disorders) | 34 (34) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No